CLINICAL TRIAL: NCT07303673
Title: Coblation Assisted Dilatation Versus Modified Maddern Procedure in Subglottic and Cervical Tracheal Stenosis: a Randomized Clinical Trial
Brief Title: Coblation Assisted Dilatation Versus Modified Maddern Procedure in Subglottic and Cervical Tracheal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD.24.05.858
Record Dates: First submitted 2025-12-07; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Subglottic Stenosis (SGS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coblation-assisted dilatation group (Active Comparator)
  Interventions: Procedure: Coblation-assisted dilatation
- Modified Maddern procedure group (Active Comparator)
  Interventions: Procedure: Modified Maddern procedure

INTERVENTIONS:
Procedure: Coblation-assisted dilatation — endoscopic Coblation-assisted dilatation is done for subglottic and / or upper tracheal stenosis. Radial incisions are done using the coblation technique, followed by balloon dilatation.
  Arms: Coblation-assisted dilatation group
Procedure: Modified Maddern procedure — endoscopic excision of the scar tissue is done in patients with subglottic and / or upper tracheal stenosis. The resultant raw surface is covered with a buccal mucosal graft harvested from the patient cheek mucosa. The donor site is closed by primary suturing.
  Arms: Modified Maddern procedure group

SUMMARY:
This study compares the effectiveness of Coblation-assisted endoscopic airway dilatation with the modified Maddern procedure-which involves endoscopic excision of scar tissue followed by buccal mucosal grafting-in patients with subglottic and/or upper tracheal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with (grade II, III) subglottic and/or upper tracheal stenosis according to Myer-Cotton grading system
* all age groups (children and adults)

Exclusion Criteria:

* Patients with cervical spine diseases where an extended position during the procedure could be problematic.
* Previous neck or oral cavity irradiation.
* chronic uncontrolled debilitating diseases that might interfere with the healing process e.g. (diabetes mellitus, renal failure, decompensated liver diseases).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Airway diameter | 3, 6, and 12 weeks
  assessment of the diameter of the airway after the procedure by endoscopic examination

SECONDARY OUTCOMES:
subjective evaluation of breathing | 3, 6, and 12 months
  the breathing is evaluated subjectively using the dyspnea handicap index. The Dyspnea Handicap Index (DHI) is a validated self-reported questionnaire consisting of 10 items, each scored as 0 (never), 2 (sometimes), or 4 (always), yielding a total score from 0 to 40, with higher scores indicating greater severity of dyspnea-related functional and emotional handicap.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kavookjian, H., & Hillel, A. (2023). Endoscopic laryngotracheoplasty (Maddern procedure) for idiopathic subglottic stenosis. Operative Techniques in Otolaryngology-Head and Neck Surgery, 34(2), 115-119.
- [Result] Pasick LJ, Anis MM, Rosow DE. An Updated Review of Subglottic Stenosis: Etiology, Evaluation, and Management. Curr Pulmonol Rep. 2022;11(2):29-38. doi: 10.1007/s13665-022-00286-6. Epub 2022 Mar 3. PMID 35261874
- [Result] Wijermars LGM, Hoekstra CEL, Nguyen TTT, Stevens MF, Dikkers FG. New Treatment Strategy for Subglottic Stenosis Using the Trachealator, a Novel Non-occlusive Balloon. Laryngoscope. 2022 Nov;132(11):2202-2205. doi: 10.1002/lary.30234. Epub 2022 May 30. No abstract available. PMID 35634800
- [Result] Lorenz RR. The Evolution and Outcomes of the "Maddern Procedure" for the Treatment of Subglottic Stenosis. Laryngoscope. 2023 Nov;133(11):3100-3108. doi: 10.1002/lary.30752. Epub 2023 May 17. PMID 37194674